CLINICAL TRIAL: NCT04807855
Title: Custom Print Megnetic Levator Prosthesis Pilot Comparison
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Skelmet Inc (Industry)
Collaborators: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Skelmet
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Blepharoptosis
Keywords: Blepharoptosis
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- the experimental arm (Experimental): All subjects, the ptosis group and the normal group receive the same intervention.
  Interventions: Device: The cMLP device

INTERVENTIONS:
Device: The cMLP device — There is only one medical device we are testing, so only one intervention.

SUMMARY:
Study the device feasibility of non-surgical treatment for blepharoptosis (inability to open the eyelid) consisting of a biocompatible magnetic element adhered to the upper eyelid and a second magnet above the eye on a custom 3D-printed eyeglasses frame with a dial to provide adjustable magnetic force to open the eye while still allowing eye closure.

DETAILED DESCRIPTION:
Extensive description of the study protocol is provided in the Research Strategy (R), but key components are summarized and justified here. This is a prospective, interventional, single-arm, single-group open label study. Because the primary objective of this study is to perform prototyping in the interest of developing and determining the feasibility of our novel approach, randomization to treatment or control is not necessary or appropriate at this stage. All participants will have ptosis and will be fitted with the experimental custom adjustable force MLP. Determining if the custom MLP is superior to the non-custom MLP is beyond the scope of this phase I SBIR project.

The primary outcome is custom MLP fitting success defined as 8mm interpalpebral fissure size or greater, patient desire to engage in a 20-min trial, and comfort rated greater than 5 out of 10 after the 20 minute trial (all criteria must be met). These criteria may be met at any one visit in the prototyping process. Therefore, one prototype may fail but if subsequent prototypes succeed, the case will be rated as a success. Selection of the criteria was based on a desire to have both objective and subjective metrics. Eye opening of 8mm was selected because it is a functional amount of eye opening found to be useful to patients in prior studies (note that these patients do not have inferior lid malposition). We have used interpalpebral fissure as a primary outcome as opposed to Marginal Reflex Distance (distance from the corneal reflection to upper lid) in order to allow enrollment of bilateral and severe cases, and to provide a common outcome for both eye opening and closing on the blink. Desire to engage in a 20-minute trial was selected as a criteria because it provides some information on the patient's opinion of the device. Comfort greater than 5 out of 10 indicates better than neutral, and was selected as a minimum goal for success (median comfort in our prior study was 8 out of 10).

The statistical analysis method for the primary outcome will be an exact binomial test of one proportion to determine which condition is met for more than half of patients. If the prototype approach is successful for greater than half of patients after 20 minutes of wear there will be a large enough sample for a phase II study to warrant continued development.

Sample Size Calculation for primary outcome: With 10 subjects we will have 80% power to show that the success rate significantly exceeds 50% with a one-sided alpha=0.05 exact binomial test of one proportion when the success rate is 8/10 or greater, meaning 8 would have to succeed to reach significance. With 15 subjects the success rate would need to be 11 to reach significance.

ELIGIBILITY:
Inclusion Criteria:

* Presence of Blepharoptosis for at least one eye, moderate cognitive function or better defined as greater than or equal to 18 out of 30 on a pre-screening of the Mini-Mental State Exam, age 5 or older. Sex - All. Gender Based - All.

Exclusion Criteria:

* Absence of Blepharoptosis. Age less than 5, Severe Cognitive impairment defined as Mini-mental score less than 18, behaviors consistent with delirium (combinations of disorientation, hallucinations, delusions, and incoherent speech), or lethargy. These individuals must be excluded since participation requires competent self-care, reliable responses and cooperation during fitting of the devices. Healthy Volunteers.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Resting interpalpebral fissure size | after 20 minutes of wear
  Interpalpebral fissure is defined as the greatest distance between the upper and lower eye lid margins at the insertion point of the lashes. Resting is defined as point where the eyelid is maximally elevated.
Patient decision to participate in a 20-min trial with the prototype MLP | after 2 minutes of wear
  This is a binary response measure (1 = yes I would like to participate or 0 = no I would not like to participate.
Comfort rating scale | after 20 minutes of wear
  This measure is a 10 point likert-type rating scale used to quantify the comfort of the MLP (1 poor comfort to 10 high comfort).

SECONDARY OUTCOMES:
Difference in the resting interpalpebral fissure size from highest to lowest magnetic force settings | after 2 minutes of wear
  Interpalpebral fissure is defined as the greatest distance between the upper and lower eye lid margins at the insertion point of the lashes. Resting is defined as point where the eyelid is maximally elevated.
Interpalpebral fissure size at maximum blink | after 2 minutes, 20 minutes, and 1-week of wear
  Interpalpebral fissure is defined as the greatest distance between the upper and lower eye lid margins at the insertion point of the lashes. Maximum blink is the point of smallest interpalpebral fissure (most closing).
Frequency and severity of adverse events | after 20 minutes and 1-week of wear
  Thresholds for adverse events include eyelid skin erythema greater than grade II on the industry scale, grade II worsening in corneal staining on the NEI industry scale, and a greater than 2-line worsening in visual acuity in the treated eye.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Cao, Mr, Principal Investigator — Skelmet Inc
Locations (1):
- Mass. Eye and Ear, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
We will not be sharing IPD with other researchers.